CLINICAL TRIAL: NCT02971189
Title: Librata Endometrial Ablation Device Treatment to Reduce Menstrual Blood Loss in Sites Across the United Kingdom
Acronym: LEADERUK
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Birmingham Women's NHS Foundation Trust (Other Government)
Responsible Party: Principal Investigator, Mr.Justin Clark, Consultant Gynaecologist, Birmingham Women's NHS Foundation Trust
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Birmingham WHC
Record Dates: First submitted 2016-11-19; First posted 2016-11-22 (Estimated); Last update posted 2016-11-22 (Estimated); Status verified 2016-11

CONDITIONS: Heavy Menstrual Bleeding
MeSH Terms: conditions — Menorrhagia

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Librata endometrial ablation (Other): Librata thermal balloon endometrial ablation treatment procedure will be performed in accordance with the physician's routine endometrial ablation practice and in accordance with the requirements of the LibrataTM IFU. The uterine cavity will be systematically inspected using hysteroscopy prior the ablative procedure (after any blind cervical dilatation) and post the ablative procedure to estimate the completeness of endometrial destruction and to exclude uterine trauma including uterine perforation. The patient will undergo standard post-operative monitoring and recovery according to usual hospital practices. An assessment will be made for any ablation procedure or device related serious adverse events.
  Interventions: Device: Librata Endometrial Ablation

INTERVENTIONS:
Device: Librata Endometrial Ablation — The treatment procedure will be performed in accordance with the physician's routine endometrial ablation practice and in accordance with the requirements of the LibrataTM IFU. The uterine cavity will be systematically inspected using hysteroscopy prior the ablative procedure (after any blind cervical dilatation) and post the ablative procedure to estimate the completeness of endometrial destruction and to exclude uterine trauma including uterine perforation. The patient will undergo standard post-operative monitoring and recovery according to usual hospital practices. An assessment will be made for any ablation procedure or device related serious adverse events.

SUMMARY:
A prospective, single-arm, non-randomised study to evaluate the Librata device performance and acute safety in performing global endometrial ablation in pre-menopausal women with heavy menstrual bleeding.

DETAILED DESCRIPTION:
4 clinical sits around the UK aim to recruit 40 women into a study to assess the primary objective of procedure success using the Librata endometrial ablation device, as defined as device success (completion of treatment cycles according to device specifications) and no occurrence of intra-procedural complications.

The investigators will also assess the secondary objectives of:

1. Rates of bleeding at months 3, 6 and 12 as measured by menstrual pictogram
2. Rate of serious adverse device effects through to day 30 post-operatively
3. Rates of re-intervention for menstrual related bleeding or pain and/or hysterectomy at 6 and 12 months
4. Rates of patient satisfaction at 6 and 12 months.

ELIGIBILITY:
Inclusion Criteria:

1. Refractory heavy menstrual bleeding with no definable organic cause
2. Female subject from (and including) age 25 to 50 years
3. Uterine sound measurement between 6.0 to 10.0cm (external os to fundus).
4. A minimum menstrual blood loss of

   * Menstrual Pictogram (MP) score of ≥150 for 3 consecutive months prior to study enrollment; OR,
   * MP score ≥150 for one month for women who either had:

     * at least 3 prior months documented failed medical therapy; or
     * a contraindication to medical therapy; or
     * refused medical therapy
5. Premenopausal at enrollment as determined by FSH measurement ≤ 40 IU/L
6. Not pregnant and no desire to conceive at any time
7. Subject agrees to use a reliable form of contraception. If a hormonal birth control method is used, the subject must have been on said method for ≥ 3 months prior to enrollment and agrees to remain on the same hormonal regimen through their study participation.
8. Able to provide written informed consent using a form that has been approved by the reviewing IRB/EC
9. Subject agrees to follow-up schedule and data collection requirements
10. Subject is literate or demonstrates an understanding on how to collect menstrual blood loss products, and use of the Menstrual Pictogram (MP) diary

Exclusion Criteria:

Participants who have or meet any of the following exclusion criteria will not be enrolled in the Study:

1. Pregnancy or subject with a desire to become pregnant
2. Endometrial hyperplasia as confirmed by histology
3. Presence of active endometritis
4. Active pelvic inflammatory disease
5. Active sexually transmitted disease (STD), at the time of ablation.

   * Note: Treatment of STD documented in the chart serves as sufficient evidence of infection resolution. Subject may be considered for study enrollment.
6. Presence of bacteraemia, sepsis, or other active systemic infection
7. Active infection of the genitals, vagina, cervix, uterus or urinary tract at the time of the procedure
8. Known/suspected gynecological malignancy within the past 5 years
9. Known clotting defects or bleeding disorders
10. Untreated/unevaluated cervical dyskaryosis (except CIN I)
11. Known or suspected abdominal/pelvic cancer
12. Prior uterine surgery (except lower segment caesarean section) that interrupts the integrity of the uterine wall (e.g., myomectomy or classical cesarean section)
13. Previous endometrial ablation procedure
14. Currently on medications that could thin the myometrial muscle, such as long-term steroid use (except inhaler or nasal therapy for asthma)
15. Currently on anticoagulants
16. Abnormal shaped uterine cavity as confirmed by transvaginal ultrasound scan +/- hysteroscopy - specifically:

    * Septate or bicornuate uterus or other congenital malformation of the uterine cavity
    * Submucosal fibroids (grade 0-2) which protrude >1cm into the uterine cavity
    * Polyps > 2cm in maximum diameter
    * Intramural or subserosal fibroid greater than 3 cm
17. Presence of an intrauterine device (IUD) which the subject unwilling to have removed at the time of the operative visit
18. Presence of an implantable contraceptive device (e.g. Essure or Adiana).
19. Subject not currently on hormonal birth control therapy and unwilling to use a non-hormonal birth control post-ablation.
20. Subject wanting concomitant hysteroscopic sterilization.
21. Subject who is within 6-weeks post-partum.
22. Any general health condition which, in the opinion of the Investigator, could represent an increased risk for the subject
23. Any subject who is currently participating or considers future participation in any other

Ages: 25 Years to 50 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 40 (Estimated)
Dates: Start 2016-12; Primary Completion 2017-01 (Estimated); Study Completion 2017-08 (Estimated)

PRIMARY OUTCOMES:
Procedure success defined as device success (completion of treatment cycles according to device specifications) and no occurence of intra-procedural complications. | Day of surgery

SECONDARY OUTCOMES:
rates of bleeding as measured by menstrual pictogram | 12 months
rate of serious adverse device effects | day 30 post-operatively
Rates of re-intervention for menstrual related bleeding or pain and/or hysterectomy | 12 months
Rates of patient satisfaction | 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Justin Clark, MB ChB, MD, Principal Investigator — Birmingham Women's NHS Foundation Trust

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Shaw RW, Brickley MR, Evans L, Edwards MJ. Perceptions of women on the impact of menorrhagia on their health using multi-attribute utility assessment. Br J Obstet Gynaecol. 1998 Nov;105(11):1155-9. doi: 10.1111/j.1471-0528.1998.tb09968.x. PMID 9853763
- See also: link to pubmed — https://www.ncbi.nlm.nih.gov/pubmed/?term=shaw+r+and+1998+and+menorrhagia